CLINICAL TRIAL: NCT00400816
Title: Phase II Trial of Continuous Dose Temozolomide in Patients With Newly Diagnosed Pure and Mixed Anaplastic Oligodendroglioma
Brief Title: Temozolomide in Treating Patients With Newly Diagnosed Anaplastic Oligodendroglioma or Mixed Oligoastrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-4204; P30CA043703 (NIH)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-01

CONDITIONS: Central Nervous System Tumors; Brain Tumor
Keywords: adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Oligodendroglioma; Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): Temozolomide, 150 mg/m2/d x days 1-7 and 15-21
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — Schedule of Temozolomide administration: Temozolomide, 150 mg/m2/d x days 1-7 and 15-21, given every 28 days [i.e., 7 days on/7 days off]
  Other Names: Temodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with newly diagnosed anaplastic oligodendroglioma or mixed oligoastrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine progression-free survival of patients with newly diagnosed anaplastic oligodendroglioma (AO) or mixed oligoastrocytoma (MOA) treated with temozolomide.
* Determine the response rate in these patients.
* Assess the quality of life of patients with AO or MOA treated with this regimen.

OUTLINE: This is a parallel-group, multicenter study. Patients are stratified according to disease type (anaplastic oligodendroglioma vs mixed oligoastrocytoma).

Patients receive oral temozolomide once daily on days 1-7 and 15-21. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before courses 1, 3, 5, and 7, every 3 months for the first year after completion of treatment, every 4 months for the second year, every 6 months for the third and fourth years, and once a year thereafter.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed anaplastic oligodendroglioma or mixed oligoastrocytoma meeting 1 of the following criteria:

  * Bidimensionally measurable disease
  * Evaluable disease
  * Nonevaluable disease as demonstrated by gross total surgical resection
* No immediate need for cranial irradiation

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,500/mm³
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.0 times ULN
* AST ≤ 3.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No infection requiring systemic antibiotics within the past 14 days
* No other malignancy within the past 5 years except for carcinoma in situ of the cervix or nonmelanoma skin cancer
* No unrelated medical problems that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for this malignancy
* No prior radiotherapy to the brain
* No surgery requiring general anesthesia > 2 hours in duration within the past 10 days
* No prior temozolomide
* Concurrent steroids allowed provided dose is stable or decreasing for at least 1 week prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01-17 (Actual); Study Completion 2016-01-06 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | Survival of Last Patient
  Time in months to patient's disease progresses

SECONDARY OUTCOMES:
Toxicity--Count of Related Advers Events | Post-Treatment
  Count of Treatment Related Toxicities

CONTACTS AND LOCATIONS:
Overall Officials: David M. Peereboom, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States